CLINICAL TRIAL: NCT04567043
Title: Reating Opioid Misuse Via Mindfulness-Based Just-in-Time Adaptive Intervention
Brief Title: Treating Opioid Misuse Via Mindfulness-Based Just-in-Time Adaptive Intervention
Acronym: MORE-JITAI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Eric Garland, Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00078615.2
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Oriented Recovery Enhancement+JITAI (Experimental): Participants will attend a telehealth Mindfulness-Oriented Recovery Enhancement (MORE) group plus mindfulness JITAI weekly for eight weeks.
  Interventions: Behavioral: MORE+JITAI
- Supportive Psychotherapy (Active Comparator): Participants will attend a telehealth supportive psychotherapy group weekly for eight weeks.
  Interventions: Behavioral: Supporive Psychotherapy

INTERVENTIONS:
Behavioral: MORE+JITAI — Mindfulness-Oriented Recovery Enhancement (MORE) is a group behavioral intervention that unites mindfulness training, cognitive reappraisal, and positive psychological principles into an integrative intervention strategy targeting mechanisms of pain and opioid misuse. JITAI involves stress-triggered reminders to practice mindfulness skills.
  Arms: Mindfulness-Oriented Recovery Enhancement+JITAI
Behavioral: Supporive Psychotherapy — A supportive psychotherapy group will allow participants to express emotions, share experiences, and receive social support under the guidance of a skilled therapist.
  Arms: Supportive Psychotherapy

SUMMARY:
This pilot RCT will examine the preliminary efficacy of a telehealth version of Mindfulness-Oriented Recovery Enhancement (MORE) enriched with a smartphone-based just-in-time adaptive intervention (JITAI) for patients with chronic pain on long-term opioid therapy.

ELIGIBILITY:
Inclusion Criteria:

* Current chronic pain diagnosis determined by physician assessment (including but not limited to ICD-9 diagnoses 338.0, 338.21, 338.22, 338.28, 338.29, 338.4)
* Current use of prescription opioid agonist or mixed agonist-antagonist analgesics for >90 days
* Willingness to participate in study interventions and assessments

Exclusion Criteria:

* Prior experience with Mindfulness-Based Stress Reduction, Mindfulness-Based Cognitive Therapy, or Mindfulness-Based Relapse Prevention
* Active suicidality, schizophrenia, psychotic disorder
* Presence of clinically unstable systemic illness judged to interfere with treatment
* No access to internet (which will prevent telehealth-based treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Change in momentary craving | Baseline through 1-month follow-up
  Craving measured by numeric rating scale via ecological momentary assessments (min 0, max 10, with higher scores meaning more craving)
Change in momentary pain: numeric rating scale | Baseline through 1-month follow-up
  Pain measured by numeric rating scale via ecological momentary assessments (min 0, max 10, with higher scores meaning more pain)

SECONDARY OUTCOMES:
Change in momentary positive affect | Baseline through 1-month follow-up
  Positive affect measured by numeric rating scale via ecological momentary assessments (min 0, max 10, with higher scores meaning more positive affect)
Change in momentary stress | Baseline through 1-month follow-up
  Stress measured by numeric rating scale via ecological momentary assessments (min 0, max 10, with higher scores meaning more stress)
Change in heart rate variability | Baseline through 1-month follow-up
  Changes in heart rate variability (HRV) measured via ambulatory HRV assessment

OTHER OUTCOMES:
Change in opioid misuse | Baseline through post-treatment (week 8)
  Scores on Current Opioid Misuse Measure, with higher scores indicating higher opioid misuse (min 0, max 68)
Change in chronic pain symptoms | Baseline through post-treatment (week 8)
  Scores on Brief Pain Inventory, with higher scores indicating higher pain severity (min 0, max 10)
Change in opioid dose | Baseline through post-treatment (week 8)
  Opioid dose as assessed with Timeline Followback Procedure
Change in self-transcendence | Baseline through post-treatment (week 8)
  Self-transcendence measured by Nondual Awareness Dimensional Assessment, with higher scores indicating higher self-transcendence (min 13, max 65)
Change in mindful reinterpretation of pain sensations | Baseline through post-treatment (week 8)
  Mindful reinterpretation of pain sensations measured by the Mindful Reinterpretation of Pain Sensations Scale, with higher scores indicating higher reinterpretation of pain sensations (min 0, max 45)

CONTACTS AND LOCATIONS:
Locations (1):
- Center on Mindfulness and Integrative Health Intervention Development, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garland EL, Manusov EG, Froeliger B, Kelly A, Williams JM, Howard MO. Mindfulness-oriented recovery enhancement for chronic pain and prescription opioid misuse: results from an early-stage randomized controlled trial. J Consult Clin Psychol. 2014 Jun;82(3):448-459. doi: 10.1037/a0035798. Epub 2014 Feb 3. PMID 24491075
- [Derived] Garland EL, Gullapalli BT, Prince KC, Hanley AW, Sanyer M, Tuomenoksa M, Rahman T. Zoom-Based Mindfulness-Oriented Recovery Enhancement Plus Just-in-Time Mindfulness Practice Triggered by Wearable Sensors for Opioid Craving and Chronic Pain. Mindfulness (N Y). 2023 May 24:1-17. doi: 10.1007/s12671-023-02137-0. Online ahead of print. PMID 37362184